CLINICAL TRIAL: NCT01175993
Title: Effects of Rapid-Resisted Exercise on Ambulatory Adults With Traumatic Brain Injury
Brief Title: Effects of Rapid-Resisted Exercise and Bright Light Therapy on Ambulatory Adults With Traumatic Brain Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100150; 10-CC-0150
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-08-08

CONDITIONS: Adult; Traumatic Brain Injury; fMRI
Keywords: Motor Training; Post-Traumatic Stress Disorder (PTSD); Balance
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eliptical training (Active Comparator): Home base exercise
  Interventions: Other: Elliptical exercise

INTERVENTIONS:
Other: Elliptical exercise — Each participant with TBI will participate in an exercise intervention which will be done in the home. The exercise device in this protocol will be an elliptical trainer that requires coordinated reciprocal movements of both the legs and the arms. Primary emphasis will be placed on maintaining a near maximal speed of movement and to progressively increase this over time. Mild resistance to the leg motion will be provided initially and will be progressively increased once speed and coordination are optimized. The device will be loaned to them to use in the home, and will be delivered to the home fully assembled. Participants will be monitored by phone the first week and thereafter every two weeks and progressed as indicated. The exercise program will be performed 5 days a week for 30 minutes per session, for a total duration of 12 weeks. All will record the length, speed and resistance of each session on a paper-based log sheet.

SUMMARY:
Background:

* Traumatic brain injury may have a range of effects, from severe and permanent disability to more subtle functional and cognitive deficits that often go undetected during initial treatment. To improve treatments and therapies and to provide a uniform quality of care, more research is needed into different treatments for traumatic brain injury.
* Exercise has been shown to improve movement and balance in people with strokes, cerebral palsy, and other conditions that affect the brain, and can improve symptoms of memory problems or depression. Bright light therapy has also been shown to improve mood in people with depression. Researchers are interested in studying problems with movement, balance, thinking, and mood in people with traumatic brain injury. By comparing the effects of exercise and bright light exposure on brain function, new treatments may be developed for acute traumatic brain injury.

Objectives:

- To compare the effects of exercise and bright light therapy on the brain function of individuals with traumatic brain injury.

Eligibility:

- Individuals between 18 and 44 years of age who either have been diagnosed with traumatic brain injury or are healthy volunteers.

Design:

* Individuals with traumatic brain injury will have four outpatient evaluation visits at the clinical center, a 3-month home exercise program, and a 3-month bright light exposure program at home. Healthy volunteers will have one evaluation visit at the clinical center.
* At the first study visit, all participants will have a full physical examination and medical history. Individuals with traumatic brain injury will also have an eye exam to determine if it is safe for them to receive light therapy.
* All participants will have the following initial tests:
* Tests of walking and movement, including monitoring by a physical therapist; tests to record joint movement and evaluate muscle function; tests that combine movement, thinking, and speaking; and balance and reaction time tests.
* Magnetic resonance imaging scans
* Tests of thinking and mood, including questionnaires, computerized tests, and simple action tests.
* Participants with traumatic brain injury will have separate 3-month sessions of exercise and bright light therapy, with additional evaluation visits between each 3-month session and at the end of the study. Between the 3-month sessions, participants will have 1 month with no intervention.
* Exercise sessions will involve regular workouts on an elliptical machine for 30 minutes for 5 days a week, and bright light therapy sessions will involve sitting in front of a light box for 30 minutes for 5 days a week. Participants will keep a journal to monitor the effects of the therapy.

DETAILED DESCRIPTION:
Objectives: We will: 1) compare performance of healthy volunteers and ambulatory adults with traumatic brain injury (TBI) on a range of motor, neurobehavioral and brain imaging outcomes; and 2) evaluate effects of rapid, reciprocal arm and leg exercise with an elliptical trainer on high-level motor coordination and balance, and neurobehavioral and cognitive functioning in persons with TBI. Brain connectivity and changes in connectivity in response to intervention will be quantified. We hypothesize even highly functional adults with TBI will have poorer scores on all measures than controls; exercise will lead to significant improvements in motor performance and balance,and neurobehavioral and cognitive functioncompared to an equivalent length of time during which they were not participating in training. We further hypothesize that improvements in cortical connectivity and representation will relate directly to functional ones.

Study Population: 80 adults (50 with TBI) will be recruited so that 20 with TBI and 20 healthy volunteers complete the study. Only the TBI group will receive intervention.

Design: Healthy controls with have a single assessment that includes motor, neuropsychological and brain imaging tests. Participants with TBI will have 3 visits with the same motor, neuropsychological and brain imaging tests as the healthy controls. They will perform 2 months of fast elliptical training. Assessments will occur at 0, 2, and 4 months. The exercise device will be an elliptical trainer that exercises the legs and arms with the emphasis on maintaining a fast speed. Mild resistance will be provided initially and progressively increased once speed is optimized. The training will be performed in the home 5 days per week for 30 minutes.

Outcome Measures: Performance on complex motor and balance tasks will be assessed with 3D motion capture & EMG, the Smart Balance Measurement System and the High Level Mobility Assessment Tool (Hi-MAT). Primary outcomes are Hi-MAT score, reaction time during balance testing and the Hamilton Rating Scale for Depression (Ham-D). Secondary outcomes will include measures of motor speed and reaction time, dual task performance, memory, anxiety, sleep quality, and responses to stress. Cortical connectivity will be quantified using resting state functional connectivity magnetic resonance imaging (MRI) and Diffusion Tensor Imaging (DTI), which evaluates white matter tracts. Cortical activation patterns during imagined walking will be quantified with fMRI.

ELIGIBILITY:
* INLCUSION CRITERIA:

Inclusion criteria for all subjects (healthy volunteers and those with TBI) include:

-ages 18 - 44, inclusive

Additional inclusion criteria for those with TBI include:diagnosis of traumatic brain injury

* at least 6 months from initial brain injury
* ability to stand and walk independently and safely without assistance
* sufficient attention and cognition to complete the assessments without a proxy
* capable of providing own consent

EXCLUSION CRITERIA:

* presence of an injury to any extremity, or other medical condition that would affect motor function or the ability to perform the assessments or the exercise program, specifically balance problems due to Vestibulopathy, that would affect your ability to perform the assessments or the exercise program
* have any of the following contraindications to having an MRI scan:

  * Pregnancy: For any female of childbearing potential who is not pregnant, a pregnancy test will be done.
  * A ventriculo-peritoneal shunt
  * Have claustrophobia and are not comfortable in small enclosed spaces.
  * have metal in your body that would make having an MRI scan unsafe such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear or ear implant, transdermal medication patch (nitroglycerine), any metallic implants or objects, body piercing that cannot be removed, bone or joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal embedded (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near your eyes). If you have a question about any metal objects being present in your body, you should ask the study doctor.
  * Excessive startle reaction to or fear of loud noises
  * You are not able to fit in the scanner

Additional exclusion criteria for those with TBI include:

-Planning to make a change in medication or therapy during the enrollment period with the goal of improving mood, cognitive function or motor function.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2014-02-04 (Actual)

PRIMARY OUTCOMES:
1. HiMAT is a composite measure of high functioning mobility skills. 2. Limits of Stability instrumented balance test wih a focus on response speed3. Hamilton Depression (HAM-D) inventory to evaluate changesin emotional health | 0, 2, and 4 months
  Primary outcomes are Hi-MAT score, reaction time during balance testing and the Hamilton Rating Scale for Depression (Ham-D).

SECONDARY OUTCOMES:
1. movement speed and reaction time during a range of motor tasks2. Other aspects of balance tests (e.g. directionality)3. scores on neuropsychological tests4. analysis of brain pathway volume and connectivity | 0, 2, and 4 months
  Secondary outcomes will include measures of motor speed and reaction time, dual task performance, memory, anxiety, sleep quality, and responses to stress. Cortical connectivity will be quantified using resting state functional connectivity magnetic resonance imaging (MRI) and Diffusion Tensor Imaging (DTI), which evaluates white matter tracts. Cortical activation patterns during imagined walking will be quantified with fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Silvina G Horovitz, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Martin EM, Lu WC, Helmick K, French L, Warden DL. Traumatic brain injuries sustained in the Afghanistan and Iraq wars. J Trauma Nurs. 2008 Jul-Sep;15(3):94-9; quiz 100-1. doi: 10.1097/01.JTN.0000337149.29549.28. PMID 18820555
- [Background] Brown AW, Elovic EP, Kothari S, Flanagan SR, Kwasnica C. Congenital and acquired brain injury. 1. Epidemiology, pathophysiology, prognostication, innovative treatments, and prevention. Arch Phys Med Rehabil. 2008 Mar;89(3 Suppl 1):S3-8. doi: 10.1016/j.apmr.2007.12.001. PMID 18295647
- [Background] Katz DI, White DK, Alexander MP, Klein RB. Recovery of ambulation after traumatic brain injury. Arch Phys Med Rehabil. 2004 Jun;85(6):865-9. doi: 10.1016/j.apmr.2003.11.020. PMID 15179637
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0150.html